CLINICAL TRIAL: NCT00750399
Title: An Open Label Study to Evaluate the Effect of Intravitreal Ranibizumab on Radiation Retinopathy Following Plaque Brachytherapy for Choroidal Melanoma
Brief Title: Effect of Intravitreal Ranibizumab on Radiation Retinopathy Following Plaque Brachytherapy for Choroidal Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The New York Eye Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Paul T. Finger, MD, Director, The New York Eye Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF4519s
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Radiation Retinopathy; Choroidal Melanoma
Keywords: radiation; retinopathy; ranibizumab; melanoma; choroid
MeSH Terms: conditions — Uveal Melanoma; Retinal Diseases; Melanoma | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravitreal ranibizumab (Experimental): Patients will receive intravitreal ranibizumab on a monthly basis depending on response to treatment
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — intravitreal ranibizumab monthly for 4 months, and then every month thereafter until month 12.
  Other Names: Lucentis
Drug: ranibizumab — intravitreal ranibizumab 0.5 mg
  Other Names: Lucentis

SUMMARY:
This is a Phase I clinical trial to test the safety and tolerability of intravitreal ranibizumab in the treatment of radiation retinopathy following plaque brachytherapy for patients with choroidal melanoma using the incidence and severity of events criteria.

The secondary objective is to assess the efficacy of intravitreal ranibizumab on regression of radiation retinopathy by ophthalmic examination, fundus photography, fluorescein angiography, and optical coherence tomography, as well as visual acuity.

DETAILED DESCRIPTION:
Following plaque brachytherapy as treatment for choroidal melanoma, patients may develop radiation retinopathy. Radiation retinopathy is a progressive condition that leads to blindness in over 50% of cases within 5 years of treatment.

Vascular endothelial growth factor (VEGF) protein is believed to play a critical role in angiogenesis and radiation retinopathy. It is one of the key contributors to physiological or pathological conditions that can stimulate both the formation of new blood vessels and normal vessel incompetence. Ranibizumab is a recently approved vascular endothelial growth factor (VEGF) inhibitor shown to be effective in treating exudative macular degeneration. Ranibizumab binds to and inhibits vascular endothelial growth factor A (VEGF-A), which has been shown to cause neovascularization and leakage in models of ocular angiogenesis.

This is an open label, non-randomized active treatment, Phase I trial to assess the safety and tolerability of intravitreal ranibizumab and its ability to reduce radiation retinopathy and potentially limit vision loss associated with this disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of radiation retinopathy
* History of choroidal melanoma status post plaque brachytherapy
* Age > 21 years
* Ability to perform written consent and comply with study assessments for the full duration of the study

Exclusion Criteria:

* Pregnancy or lactation, pre-menopausal women not using contraception
* Participation in another simultaneous medical investigation or trial
* Patient with significantly compromised visual acuity in the study eye due to concomitant ocular conditions.
* Patients who have undergone intraocular surgery within last 60 days.
* Patients who have had intravitreal anti-VEGF treatment within 45 days.
* Patients who have had intravitreal triamcinolone acetonide within 4 months.
* Patients who have had laser within 60 days.
* Inability to obtain photographs to document CNV (including difficulty with venous access).
* Patient has a history of any medical condition which would preclude scheduled visits or completion of study.
* Aphakia or absence of the posterior capsule in the study eye. Previous violation of the posterior capsule in the study eye is also excluded unless as a result of yttrium aluminum garnet (YAG) posterior capsulotomy in association with posterior chamber lens implantation..
* History of glaucoma filtering surgery in the study eye.
* Concurrent use of more than two therapies for glaucoma.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To test the safety and tolerability of intravitreal ranibizumab in the treatment of radiation retinopathy associated with plaque brachytherapy for choroidal melanoma | 12 months

SECONDARY OUTCOMES:
To assess the efficacy of intravitreal ranibizumab on treating radiation retinopathy following plaque brachytherapy for choroidal melanoma, and effect on visual acuity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul T Finger, MD, Principal Investigator — The New York Eye Cancer Center
Locations (1):
- The New York Eye Cancer Center, New York, New York, United States

REFERENCES:
- [Background] Finger PT. Radiation retinopathy is treatable with anti-vascular endothelial growth factor bevacizumab (Avastin). Int J Radiat Oncol Biol Phys. 2008 Mar 15;70(4):974-7. doi: 10.1016/j.ijrobp.2007.11.045. PMID 18313522
- [Background] Finger PT, Chin K. Anti-vascular endothelial growth factor bevacizumab (avastin) for radiation retinopathy. Arch Ophthalmol. 2007 Jun;125(6):751-6. doi: 10.1001/archopht.125.6.751. PMID 17562985
- [Result] Finger PT, Chin KJ. Intravitreous ranibizumab (lucentis) for radiation maculopathy. Arch Ophthalmol. 2010 Feb;128(2):249-52. doi: 10.1001/archophthalmol.2009.376. No abstract available. PMID 20142553